CLINICAL TRIAL: NCT03422328
Title: mUlticenter, Single-arM, Open-laBel, Long-teRm Safety Study With macitEntan in Patients With puLmonary Arterial Hypertension previousLy Treated With mAcitentan in Clinical Studies
Brief Title: A Clinical Study to Investigate the Long-term Safety of the Drug Macitentan in Patients With Pulmonary Hypertension Who Were Previously Treated With Macitentan in Clinical Studies.
Acronym: UMBRELLA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-314; 2017-003934-10 (EudraCT Number)
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension
Keywords: macitentan; long-term safety; open-label; single-arm
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Intervention Model Description: The study is designed as an open-label, single-arm, multicenter trial in which all participants roll over from a "parent study" in order to continue their dose of macitentan 10 mg once every day as already received in the "parent study".
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label macitentan 10 mg (Experimental): 10 mg macitentan film coated tablet, administered orally once daily
  Interventions: Drug: macitentan

INTERVENTIONS:
Drug: macitentan — macitentan 10 mg, film-coated tablet, oral use
  Other Names: ACT-064992; JNJ-67896062

SUMMARY:
The aim of the trial is to study the long-term safety of macitentan and to provide continued treatment with macitentan to patients with pulmonary arterial hypertension (PAH) and Chronic thromboembolic pulmonary hypertension (CTEPH) who were previously treated with macitentan in clinical studies.

DETAILED DESCRIPTION:
The purpose of this study is to provide continued treatment with macitentan to subjects with PAH or CTEPH who participated in "parent studies" and to continue to accrue long-term safety data. The design of this study is widely used in clinical programs to give participants in a clinical study access to an effective study treatment beyond completion of the parent study. This is considered the best option to collect long-term safety and tolerability information of macitentan 10 mg and survival status of participants with PAH and CTEPH. "Parent study/studies" refer to a number of clinical studies with macitentan that are conducted in different clinical classification of PAH and CTEPH (NCT00667823, NCT02112487, NCT02310672, NCT02968901, NCT02558231, NCT02382016, NCT02060721) and may be completed before the participants have access to commercial macitentan in their country of residence. The "parent studies" are fully or partially running in countries where no access to commercial macitentan is expected in the near future.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to take part in the study before any study mandated procedure.
2. Participants from one of the parent studies and: a) the sponsor has decided to terminate the parent study in that country and b) the participant has completed the end of treatment (EOT) Visit of the parent study
3. Women of childbearing potential are able to take part in the study if the following applies: a) Urine pregnancy test is negative at Enrollment; b) Agreement to perform monthly urine or serum pregnancy tests during the study and up to at least 30 days after the study treatment discontinuation; and c) Agreement to adhere to the planned contraception scheme from Enrollment up to at least 30 days after study treatment discontinuation

Exclusion Criteria:

1. Hemoglobin less than 80 gram per liter (g/L)
2. Serum Aspartate aminotransferase (AST) and/or alanine aminotransferases (ALT) more than three times the upper limit of normal range
3. Known and documented history of severe hepatic impairment that is Child-Pugh Class C.
4. Pregnant, planning to become pregnant, or breastfeeding
5. Known hypersensitivity to macitentan, its excipients, or drugs of the same class
6. Planned or current treatment with another investigational treatment up to 3 months prior to Enrollment
7. Any known factor or disease that may interfere with treatment compliance, study conduct, or interpretation of the results, such as drug or alcohol dependence or psychiatric disease
8. Treatment with a strong CYP3A4 inhibitor (e.g., ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, and saquinavir)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Incident Rate of Treatment-emergent Adverse Event | From Day 1 to End of study (EoS) visit (an average of 3 years)
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. A treatment-emergent AE is any AE temporally associated with the use of study treatment.
Incident rate of treatment-emergent adverse events (AEs) leading to premature discontinuation of study treatment | From Day 1 to EoS visit (an average of 3 years)
  Any AE will be recorded that 1) is (temporally) associated with the use of study treatment whether or not considered by the investigator as related to study treatment and 2) leads to premature discontinuation of study medication.
Incident rate of treatment-emergent serious adverse events (SAEs) | From Day 1 to EoS visit (an average of 3 years)
  Any SAE as defined by the ICH guidelines will be recorded. Any hepatic AE that leads to discontinuation of study treatment will be defined as SAE.
Number of pregnancies with maternal exposure to macitentan | From Day 1 to EoS visit (an average of 3 years)
  Pregnancies with maternal exposure to macitentan will be recorded.

OTHER OUTCOMES:
Change of WHO functional class to each scheduled time point | From Day 1 to EoT visit (an average of 3 years)
  The proportion of patients who worsened, remain unchanged or improved from baseline to each scheduled time-point in WHO function will be calculated, where baseline is the initial baseline from the "parent study" (or the double-blind core study preceding the "parent study").
Assessment of survival status at End-of-Study (EoS) | From Day 1 to EoS visit (an average of 3 years)
  Time to death of all causes up to EoS from the date of randomization or enrollment in the "parent study" (or the double-blind core study preceding the "parent study") will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Sochor, Study Director — Actelion
Locations (34):
- The Republican Scientific-Practical Center ''Cardiology'', Minsk, Belarus
- UZ Leuven, Leuven, Belgium
- France (22):
  - CHRU Besancon Hopital Jean Minjoz, Besançon
  - CHU de Bordeaux - Hospital Haut-Leveque, Bordeaux (Pessac)
  - CHU de la Cavale Blanche, Brest
  - GH est - Hôpital Cardiovasculaire et Pneumologie Louis Pradel, Bron
  - Hôpital Côte de Nacre, Caen
  - CHU Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Hopital Bicetre Aphp Hopitaux Universitaires Paris Sud, Le Kremlin-Bicêtre
  - Hôpital Cardiologique - Chru Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de la Timone, Marseille
  - CHU de Montpellier - Arnaud de Villeneuve, Montpellier
  - CHU Nantes - Hopital Nord Laënnec, Nantes
  - Centre Hospitalier Universitaire - de Nice - Hopital Pasteur, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - CHU de Reims, Reims
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHU Rouen Hopital Charles Nicolle, Rouen
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Nouvel Hopital Civil, Strasbourg
  - Hopital Larrey CHU de Toulouse, Toulouse
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Poland (2):
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - Wojewodzki Szpital Specjalistyczny Oddzial Kardiologiczny, Wroclaw
- Russia (5):
  - Cardiovascular Pathology Research Institute of Siberian Branch of RAMS, Kemerovo
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - Federal State Budgetary Institution Of Ministry Of Health Of Russian Federation, Novosibirsk
  - Federal North-West Medical Research Centre, Saint Petersburg
  - Federal State Budget Scientific Institution, Tomsk
- Istanbul University Istanbul Medical Faculty, Capa_Istanbul, Turkey (Türkiye)
- Ukraine (2):
  - CE 'Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiosurgery', Dnipro
  - Lviv Regional Clinical Hospital, Lviv